CLINICAL TRIAL: NCT01005355
Title: Phase 1 Study of IMC-1121B in Patients With Advanced Solid Tumors
Brief Title: Study of IMC-1121B in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13898; CP12-0816 (Other: ImClone Systems); I4T-IE-JVBI (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-10-05; First posted 2009-10-30 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Solid Tumors
Keywords: Solid tumor; recombinant human IgG1; MAB; monoclonal antibody; VEGFR 2; human vascular endothelial growth factor receptor 2
MeSH Terms: interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMC-1121B (Experimental): Participants receiving IMC-1121B intravenously
  Interventions: Biological: IMC-1121B

INTERVENTIONS:
Biological: IMC-1121B — Cycle 1: Upon completion of enrollment criteria confirmed at screening, the first dose of study medication should be administered within 7 days. The infusion will be planned every 2 weeks or every 3 weeks on the same day of the week of the first infusion. Dose escalation to Cohort 2 may occur in the absence of a dose-limiting toxicity (DLT) in the first three participants treated in Cohort 1 during the initial 6-week dosing period (Cycle 1). The same procedure will be followed for dose escalation from Cohort 2 to Cohort 3. If 1 of 3 participants in any cohort experiences a DLT in the first 6 weeks (Cycle 1), 3 additional participants will be enrolled in that cohort. Dose escalation to the next cohort may occur if less that 2 of 6 participants experience a DLT during Cycle 1.
  Other Names: RAMUCIRUMAB; LY3009806

SUMMARY:
This trial is testing the investigational drug IMC-1121B administered to Japanese participants with advanced solid tumors who have not responded to standard therapy or for whom no standard therapy is available. The rationale for performing this trial is to establish the safety profile and the pharmacokinetics of IMC-1121B.

DETAILED DESCRIPTION:
This single center, open-label, single-arm, Phase 1 study will enroll approximately 15 to 18 participants. The actual size will vary depending on the dose-limiting toxicities (DLTs) observed and the resultant sizes of the cohorts. Participants will receive IMC-1121B, administered intravenously, once every 2 or 3 weeks for 6 weeks (one cycle). After one cycle of treatment, participants who have an objective response or stable disease may continue to receive IMC-1121B at the same dose and schedule until disease progression or other withdrawal criteria are met. A minimum of three participants will be enrolled in each cohort. Dose escalation in successive cohorts will occur once all participants complete one cycle of therapy.

Participants will be enrolled sequentially into each cohort.

A completed participant will be either a participant who completes the initial 6 week treatment period (Cycle 1) or a participant who discontinues therapy for an IMC-1121B related toxicity during Cycle 1. Participants who do not complete the first 6 weeks of treatment for reasons other than an IMC-1121B -related toxicity will be replaced. Toxicity data for each cohort will be reviewed prior to dose escalation. Upon completion of all required safety evaluations during the initial 6 weeks, the next cohort of new participants will be treated at the next higher dose level using a dose escalation scheme.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor participant who was been histopathologically or cytologically documented.
* Advanced primary or recurrent solid tumors participant who has not responded to standard therapy or no standard therapy is available.
* The participant has measurable or nonmeasurable lesions according to Response Evaluation Criteria in Solid Tumors (RECIST).
* The participant has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-1 at study entry.
* The participant is able to provide written informed consent.
* The participant is age 20 years or older.
* The participant has a life expectancy of > 3 months.
* The participant has adequate hematologic function, as defined by:
* An absolute neutrophil count (ANC) > 1500/cubic millimeter (mm³) or /microliter (µL)
* A hemoglobin level > 10 grams/deciliter (g/dL)
* A platelet count > 100,000/mm³ or /µL
* The participant has adequate hepatic function, as defined by:
* A total bilirubin level < 1.8 milligrams/deciliter (mg/dL)
* Aspartate transaminase (AST) levels < 86 International Units/liter (IU/L)
* Alanine transaminase (ALT) levels ≤ 86 IU/L
* The participant has adequate renal function, as defined by:
* Serum creatinine level ≤ 1.5 mg/dL, or
* Calculated serum creatinine clearance (Cockcroft-Gault) ≥ 60 milliliters/minute (mL/min)
* The participant's urinary protein is 0 on dipstick or 1+ but participant does not have edema nor serum albumin < lower level of normal (LLN).
* The participant has adequate coagulation function, as defined by international normalized ratio (INR) ≤ 1.5.
* The participant agrees to use adequate contraception during the study period and for 12 weeks after the last dose of study treatment.

Exclusion Criteria:

* The participant has had chemotherapy or therapeutic radiotherapy within 28 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or participant has ongoing side effects ≥ Grade 2 due to agents administered more than 28 days earlier.
* The participant has obvious evidence of intratumor cavitation.
* The participant has undergone major surgery (example, laparotomy, thoracotomy, removal of organ[s]) within 28 days prior to study entry, or subcutaneous venous access device placement within 7 days prior to study entry.
* The participant has a history of postoperative bleeding complications or wound complications from a surgical procedure.
* The participant has elective or planned surgery to be conducted during the trial.
* The participant has documented and/or symptomatic brain or leptomeningeal metastases. (Participants who are clinically stable [no symptoms during 4 weeks prior to the enrollment] with an assessment that no further treatment [radiation, surgical excision, and administration of steroids] is required, are permitted to enter the study.)
* The participant has uncontrolled intercurrent illness including, but not limited to:
* Thrombotic or hemorrhagic disorders
* Hemoptysis (approximately one-half of a teaspoon)
* Ongoing or active infection requiring systemic antibiotic treatment
* Congestive heart failure (Class III or IV of the New York Heart Association classification for heart disease)
* Angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
* Uncontrolled hypertension (systolic blood pressure > 150 millimeters of mercury (mmHg), diastolic blood pressure > 95 mm Hg)
* Cardiac arrhythmia requires treatment [National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3.0 (NCI-CTCAE v 3.0), Grade 3], or asymptomatic sustained ventricular tachycardia)
* Peripheral neuropathy of any etiology ≥ Grade 2 (NCI-CTCAE v 3.0)
* The participant has participated in clinical studies of non-approved experimental agents or procedures within 4 weeks prior to study entry for small molecules, or 8 weeks prior to study entry for non-approved monoclonal antibodies.
* The participant, if female, is pregnant (confirmed by urine or serum pregnancy test) or lactating.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- ImClone Investigational Site, Tokyo, Japan

REFERENCES:
- [Derived] Nokihara H, Yamamoto N, Yamada Y, Honda K, Asahina H, Tamura Y, Hozak RR, Gao L, Suzukawa K, Enatsu S, Tamura T. A phase 1 study of ramucirumab in Japanese patients with advanced solid tumors. Jpn J Clin Oncol. 2017 Apr 1;47(4):298-305. doi: 10.1093/jjco/hyx008. PMID 28158463

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A participant was considered to have completed the study if he or she completed the initial 6-week treatment period (Cycle 1) or if he or she discontinued therapy because of an IMC-1121B (ramucirumab)-related toxicity during Cycle 1.
Groups:
- IMC-1121B 6 mg/kg (Cohort 1): 6 milligrams/kilogram (mg/kg) IMC-1121B (ramucirumab) based on participant's body weight administered intravenously over 1 hour on Day 1 every 2 weeks for 6 weeks (1 cycle).
  After 1 cycle of treatment, participants who had an objective response or stable disease were permitted to receive IMC-1121B (ramucirumab) at the same dose and schedule until disease progression or unacceptable toxicity occurred, or another withdrawal criterion was met.
- IMC-1121B 8 mg/kg (Cohort 2): 8 mg/kg IMC-1121B (ramucirumab) based on participant's body weight administered intravenously over 1 hour on Day 1 every 2 weeks for 6 weeks (1 cycle).
  After 1 cycle of treatment, participants who had an objective response or stable disease were permitted to receive IMC-1121B (ramucirumab) at the same dose and schedule until disease progression or unacceptable toxicity occurred, or another withdrawal criterion was met.
- IMC-1121B 10 mg/kg (Cohort 3): 10 mg/kg IMC-1121B (ramucirumab) based on participant's body weight administered intravenously over 1 hour on Day 1 every 3 weeks for 6 weeks (1 cycle).
  After 1 cycle of treatment, participants who had an objective response or stable disease were permitted to receive IMC-1121B (ramucirumab) at the same dose and schedule until disease progression or unacceptable toxicity occurred, or another withdrawal criterion was met.
Period: Overall Study
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2) | IMC-1121B 10 mg/kg (Cohort 3)
Started | 3 | 6 | 6
Received at Least 1 Dose of Study Drug | 3 | 6 | 6
Completed | 3 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2) | IMC-1121B 10 mg/kg (Cohort 3) | Total
Number analyzed (Participants) | 3 | 6 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 4 | 13
  >=65 years | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 3 | 9
  Male | 2 | 1 | 3 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 6 | 6 | 15
Region of Enrollment [Number; unit: participants]
  Japan | 3 | 6 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-Related Adverse Events
Description: Data presented are the number of participants who experienced adverse events (AE) of any grade, AE of Grade ≥3 based on National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3.0 (NCI-CTCAE v 3.0), serious adverse events (SAE) and AE resulting in death that was considered to be related to IMC-1121B (ramucirumab). A summary of SAEs and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline to study completion up to 48 weeks
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2) | IMC-1121B 10 mg/kg (Cohort 3)
Number analyzed (Participants) | 3 | 6 | 6
participants
  AE of any grade | 3 | 6 | 6
  AE of Grade ≥3 | 0 | 0 | 1
  SAE | 0 | 0 | 1
  AE resulting in death | 0 | 0 | 0

2. Primary Outcome: IMC-1121B Pharmacokinetics: Maximum Serum Concentration (Cmax) - Cohorts 1 and 2 During Cycles 1 and 2
Time Frame: Day 1 to Day 15 of Cycles 1 and 2 of a 6-week cycle
Population: All participants in Cohorts 1 and 2 who received study drug and had sufficient pharmacokinetics data to calculate Cmax for Cycles 1 and 2.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2)
Number analyzed (Participants) | 3 | 6
micrograms/milliliter (mcg/mL)
  Cycle 1 | 284 (63.7) | 371 (113)
  Cycle 2 (n=1, 2) | 352 (NA) — Only 1 participant included in the analysis, therefore standard deviation is not calculable. | 694 (123)

3. Primary Outcome: IMC-1121B Pharmacokinetics: Maximum Serum Concentration (Cmax) - Cohorts 1 and 2 During Cycles 3 to 5
Description: Due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5, Cmax could not be calculated.
Time Frame: Cycles 3, 4 and 5 of a 6-week cycle: predose and 1 hour postdose
Population: Zero participants were analyzed due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5.
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2)
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: IMC-1121B Pharmacokinetics: Area Under the Concentration (AUC) Versus Time Curve - Cohorts 1 and 2 During Cycles 1 and 2
Description: AUC for Cycle 1 is AUC from time zero to infinity [AUC(0-∞)] and for Cycle 2 is AUC over a dosing interval (AUCτ).
Time Frame: Day 1 to Day 15 of Cycles 1 and 2 of a 6-week cycle
Population: All participants in Cohorts 1 and 2 who received study drug and had sufficient pharmacokinetics data to calculate AUC(0-∞) for Cycle 1 and AUCτ for Cycle 2.
Measure: Mean (Standard Deviation); unit: micrograms*hour/milliliter (mcg*h/mL)
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2)
Number analyzed (Participants) | 1 | 2
micrograms*hour/milliliter (mcg*h/mL)
  Cycle 1 - AUC(0-∞) (n=1, 1) | 36900 (NA) — Only 1 participant included in the analysis, therefore standard deviation is not calculable. | 73800 (NA) — Only 1 participant included in the analysis, therefore standard deviation is not calculable.
  Cycle 2 - AUCτ (n=1, 2) | 56400 (NA) — Only 1 participant included in the analysis, therefore standard deviation is not calculable. | 102000 (10400)

5. Primary Outcome: IMC-1121B Pharmacokinetics: Area Under the Concentration (AUC) - Cohorts 1 and 2 During Cycles 3 to 5
Description: Due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5, AUC could not be calculated.
Time Frame: Cycles 3, 4 and 5 of a 6-week cycle: predose and 1 hour postdose
Population: Zero participants were analyzed due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5.
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: IMC-1121B Pharmacokinetics: Half-Life (t1/2) - Cohorts 1 and 2 During Cycles 1 and 2
Time Frame: Day 1 to Day 15 of Cycles 1 and 2 of a 6-week cycle
Population: All participants in Cohorts 1 and 2 who received study drug and had sufficient pharmacokinetics data to calculate t1/2 for Cycles 1 and 2.
Measure: Median (Full Range); unit: hours
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2)
Number analyzed (Participants) | 3 | 2
hours
  Cycle 1 | 158 (NA) [129 to 166] | 165 (NA) [140 to 191]
  Cycle 2 (n=0, 0) | NA (NA) [NA to NA] — Zero participants were analyzed due to the sparse pharmacokinetic sampling schedule. | NA (NA) [NA to NA] — Zero participants were analyzed due to the sparse pharmacokinetic sampling schedule.

7. Primary Outcome: IMC-1121B Pharmacokinetics: Half-Life (t 1/2) - Cohorts 1 and 2 During Cycles 3 to 5
Description: Due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5, t1/2 could not be calculated.
Time Frame: Cycles 3, 4 and 5 of a 6-week cycle: predose and 1 hour postdose
Population: Zero participants were analyzed due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5.
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2)
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: IMC-1121B Pharmacokinetics: Steady State Volume of Distribution (Vss) - Cohorts 1 and 2 During Cycles 1 and 2
Time Frame: Day 1 to Day 15 of Cycles 1 and 2 of a 6-week cycle
Population: All participants in Cohorts 1 and 2 who received study drug and had sufficient pharmacokinetics data to calculate Vss for Cycle 1. Vss is not calculated for multiple doses, therefore zero participants were analyzed for Cycle 2.
Measure: Mean (Standard Deviation); unit: milliliters/kilogram (mL/kg)
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2)
Number analyzed (Participants) | 1 | 1
milliliters/kilogram (mL/kg)
  Cycle 1 | 25.0 (NA) — Only 1 participant included in the analysis, therefore standard deviation is not calculable. | 21.4 (NA) — Only 1 participant included in the analysis, therefore standard deviation is not calculable.
  Cycle 2 (n=0, 0) | NA (NA) — Vss is not calculated for multiple doses. | NA (NA) — Vss is not calculated for multiple doses.

9. Primary Outcome: IMC-1121B Pharmacokinetics: Steady State Volume of Distribution (Vss) - Cohorts 1 and 2 During Cycles 3 to 5
Description: Due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5, Vss could not be calculated.
Time Frame: Cycles 3, 4 and 5 of a 6-week cycle: predose and 1 hour postdose
Population: Zero participants were analyzed due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5.
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2)
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: IMC-1121B Pharmacokinetics: Maximum Serum Concentration (Cmax) - Cohort 3 During Cycles 1 and 2
Time Frame: Day 1 to Day 22 of Cycles 1 and 2 of a 6-week cycle
Population: All participants in Cohort 3 who received study drug and had sufficient pharmacokinetics data to calculate Cmax for Cycles 1 and 2.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | IMC-1121B 10 mg/kg (Cohort 3)
Number analyzed (Participants) | 6
micrograms/milliliter (mcg/mL)
  Cycle 1 | 493 (122)
  Cycle 2 (n=2) | 793 (367)

11. Primary Outcome: IMC-1121B Pharmacokinetics: Maximum Serum Concentration (Cmax) - Cohort 3 During Cycles 3 to 5
Description: Due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5, Cmax could not be calculated.
Time Frame: Cycles 3, 4 and 5 of a 6-week cycle: predose and 1 hour postdose
Population: Zero participants were analyzed due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5.
Arm/Group | IMC-1121B 10 mg/kg (Cohort 3)
Number analyzed (Participants) | 0

12. Primary Outcome: IMC-1121B Pharmacokinetics: Area Under the Concentration (AUC) - Cohort 3 During Cycles 1 and 2
Description: AUC for Cycle 1 is AUC from time zero to infinity [AUC(0-∞)] and for Cycle 2 is AUC over a dosing interval (AUCτ).
Time Frame: Day 1 to Day 22 of Cycles 1 and 2 of a 6-week cycle
Population: All participants in Cohort 3 who received study drug and had sufficient pharmacokinetics data to calculate AUC(0-∞) for Cycle 1 and AUCτ for Cycle 2.
Measure: Mean (Standard Deviation); unit: micrograms*hour/milliliter (mcg*h/mL)
Arm/Group | IMC-1121B 10 mg/kg (Cohort 3)
Number analyzed (Participants) | 2
micrograms*hour/milliliter (mcg*h/mL)
  Cycle 1 - AUC(0-∞) | 61600 (17100)
  Cycle 2 - AUCτ | 103000 (26200)

13. Primary Outcome: IMC-1121B Pharmacokinetics - Area Under the Concentration (AUC) - Cohort 3 During Cycles 3 to 5
Description: Due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5, AUC could not be calculated.
Time Frame: Cycles 3, 4 and 5 of a 6-week cycle: predose and 1 hour postdose
Population: Zero participants were analyzed due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5.
Arm/Group | IMC-1121B 10 mg/kg (Cohort 3)
Number analyzed (Participants) | 0

14. Primary Outcome: IMC-1121B Pharmacokinetics: Half-Life (t1/2) - Cohort 3 During Cycles 1 and 2
Time Frame: Day 1 to Day 22 of Cycles 1 and 2 of a 6-week cycle
Population: All participants in Cohort 3 who received study drug and had sufficient pharmacokinetics data to calculate t1/2 for Cycles 1 and 2.
Measure: Median (Full Range); unit: hours
Groups:
- IMC-1121B 10 mg/kg (Cohort 3): 10 mg/kg IMC-1121B (ramucirumab) based on participant's body weight administered intravenously over 1 hour on Day 1 every 2 weeks for 6 weeks (1 cycle).
  After 1 cycle of treatment, participants who had an objective response or stable disease were permitted to receive IMC-1121B (ramucirumab) at the same dose and schedule until disease progression or unacceptable toxicity occurred, or another withdrawal criterion was met.
Arm/Group | IMC-1121B 10 mg/kg (Cohort 3)
Number analyzed (Participants) | 3
hours
  Cycle 1 | 234 (NA) [166 to 241]
  Cycle 2 (n=1) | 329 (NA) [329 to 329]

15. Primary Outcome: IMC-1121B Pharmacokinetics: Half-Life (t 1/2) - Cohort 3 During Cycles 3 to 5
Description: Due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5, t1/2 could not be calculated.
Time Frame: Cycles 3, 4 and 5 of a 6-week cycle: predose and 1 hour postdose
Population: Zero participants were analyzed due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5.
Arm/Group | IMC-1121B 10 mg/kg (Cohort 3)
Number analyzed (Participants) | 0

16. Primary Outcome: IMC-1121B Pharmacokinetics: Steady State Volume of Distribution (Vss) - Cohort 3 During Cycles 1 and 2
Time Frame: Day 1 and Day 22 of Cycles 1 and 2 of a 6-week cycle
Population: All participants in Cohort 3 who received study drug and had sufficient pharmacokinetics data to calculate Vss for Cycle 1. Vss is not calculated for multiple doses, therefore zero participants were analyzed for Cycle 2.
Measure: Mean (Standard Deviation); unit: milliliters/kilogram (mL/kg)
Arm/Group | IMC-1121B 10 mg/kg (Cohort 3)
Number analyzed (Participants) | 2
milliliters/kilogram (mL/kg)
  Cycle 1 | 40.7 (1.22)
  Cycle 2 (n=0) | NA (NA) — Vss is not calculated for multiple doses.

17. Primary Outcome: IMC-1121B Pharmacokinetics: Steady State Volume of Distribution (Vss) - Cohort 3 During Cycles 3 to 5
Description: Due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5, Vss could not be calculated.
Time Frame: Cycles 3, 4 and 5 of a 6-week cycle: predose and 1 hour post-dose
Population: Zero participants were analyzed due to the sparse pharmacokinetic sampling employed in Cycles 3 to 5.
Groups:
- IMC-1121B 10 mg/kg: 10 mg/kg IMC-1121B (ramucirumab) based on participant's body weight administered intravenously over 1 hour on Day 1 every 3 weeks for 6 weeks (1 cycle).
  After 1 cycle of treatment, participants who had an objective response or stable disease were permitted to receive IMC-1121B (ramucirumab) at the same dose and schedule until disease progression or unacceptable toxicity occurred, or another withdrawal criterion was met.
Arm/Group | IMC-1121B 10 mg/kg
Number analyzed (Participants) | 0

18. Secondary Outcome: Screen for the Development of Circulating Antibodies Against IMC-1121B (Immunogenicity)
Description: Data presented are the number of participants with treatment emergent antibody positive.
Time Frame: Baseline to study completion up to 48 weeks
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2) | IMC-1121B 10 mg/kg (Cohort 3)
Number analyzed (Participants) | 3 | 6 | 6
participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | IMC-1121B 6 mg/kg (Cohort 1) | IMC-1121B 8 mg/kg (Cohort 2) | IMC-1121B 10 mg/kg (Cohort 3)
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/6 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-1121B 6 mg/kg (Cohort 1) (N=3) | IMC-1121B 8 mg/kg (Cohort 2) (N=6) | IMC-1121B 10 mg/kg (Cohort 3) (N=6)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IMC-1121B 6 mg/kg (Cohort 1) (N=3) | IMC-1121B 8 mg/kg (Cohort 2) (N=6) | IMC-1121B 10 mg/kg (Cohort 3) (N=6)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Myodesopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 3 (5)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 1 (5) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Blood albumin decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram T wave amplitude decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (5) | 5 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 3 (4) | 0 (0)
Breast haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/1 (3) | 0/5 (0) | 0/3 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 3 (9) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.